CLINICAL TRIAL: NCT00295516
Title: Minimally Invasive Management of Rh Alloimmunization: Can Amniotic Fluid DeltaOD450 Measurements Be Replaced by Doppler Studies?
Brief Title: Doppler or Amniocentesis to Predict Fetal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Stichting Oranjekliniek, The Netherlands (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSH-REB 01-0266-U; PSI Grant Number:01-13
Record Dates: First submitted 2006-02-22; First posted 2006-02-23 (Estimated); Last update posted 2006-05-24 (Estimated); Status verified 2006-02

CONDITIONS: Rh Isoimmunization
Keywords: Rhesus; Isoimmunization; Red Cell Alloimmunization; Fetal Hemolytic Anemia; Erythroblastosis fetalis
MeSH Terms: conditions — Erythroblastosis, Fetal

INTERVENTIONS:
Procedure: Fetal Middle Cerebral Artery Doppler measurement

SUMMARY:
In pregnancies complicated by Rhesus disease, the mother has developed antibodies which cross the placenta and can cause anemia and death of the fetus. When the anemia is detected on time, the fetus can be saved by giving it blood transfusions during the pregnancy.

The standard test to predict whether the fetus needs a blood transfusion is examination of the amniotic fluid. To obtain this fluid a needle has to be inserted in the womb, which has a risk of preterm delivery, infection, and making the disease worse. This is called amniocentesis.

A new safe test, using Doppler ultrasound, has been developed to possibly replace the amniocentesis.

The aim of this study is to compare the new Doppler test with the standard amniocentesis. If the Doppler test is at least as good, this safe test may replace the amniocentesis in the management of pregnancies with Rhesus disease.

DETAILED DESCRIPTION:
In pregnancies complicated by red cell alloimmunization, the fetus may suffer from chronic progressive hemolytic anemia. Severe fetal anemia leading to hydrops and fetal demise can occur as early as 17 weeks' gestation, while in other pregnancies the only manifestation of the disease is neonatal hyperbilirubinemia. The standard of care in the management of these pregnancies is to select patients at risk of fetal anemia using information about their obstetric history, and serial maternal serum antibody measurements. The selected patients are followed closely, usually in referral centers with a special interest and expertise in managing this now relatively rare disease. Ultrasound evaluation of fetal condition, with emphasis on signs of fetal hydrops, is performed regularly. In addition, serial amniocentesis is done to assess amniotic fluid bilirubin (deltaOD450) values. This spectrophotometric method estimates the level of bilirubin in the amniotic fluid, which correlates with the severity of the hemolytic process.

Although this diagnostic test, introduced by Liley in 1961, has served fetal medicine specialists well for almost 40 years, the invasive nature of the method is considered a serious disadvantage. Furthermore, its reliability has been questioned, especially when used in the second trimester. In the past decade, noninvasive alternative methods to predict the degree of fetal anemia have been developed.

The most promising of these new diagnostic tests is Doppler measurement of fetal blood flow velocities. Fetal blood flow velocity has been shown to correlate linearly with the degree of anemia. Recently, middle cerebral artery (MCA) peak flow velocity measurements have been reported to reliably predict presence or absence of fetal anemia.

The aim of this study is to compare the performance of this new noninvasive diagnostic test with the standard test, amniocentesis for amniotic fluid deltaOD450 values. In an international multicenter setting, a large cohort of consecutive Rh-alloimmunized pregnancies will be studied prospectively. Both diagnostic tests will be performed simultaneously in all patients, and compared with the "gold standard", fetal blood sampling (FBS) to assess the actual hemoglobin concentration.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with red cell alloimmunization associated with a risk of fetal anemia (D, E, c or Duffy (Fya )antibodies, alone or in combination with other antibodies)
* Gestational age between 12 and 34 weeks at study entry, viable fetus and accurate dating
* Maternal serum test-result, above the threshold at which the fetus is considered to be at risk of developing hemolytic anemia and thus a potential candidate for invasive testing.

Exclusion Criteria:

* Presence of Kell-antibodies
* Presence of fetal hydrops at first ultrasonographic examination
* Major fetal congenital or chromosomal anomalies

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157
Dates: Start 2000-10; Study Completion 2004-08

PRIMARY OUTCOMES:
Sensitivity Middle Cerebral Artery (MCA) peak velocity Doppler measurement and amniotic fluid deltaOD450 measurements, to predict fetal anemia requiring transfusion.
Specificity of Middle Cerebral Artery (MCA) peak velocity Doppler measurement and amniotic fluid deltaOD450 measurements, to predict fetal anemia requiring transfusion.

SECONDARY OUTCOMES:
Comparison of the sensitivity and specificity of the original, linearly extended Liley chart with the Queenan (1993) chart, by plotting the deltaOD450 results found in our study in both charts.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Oepkes, MD, PhD, Principal Investigator — Leiden University Medical Centre, The Netherlands; Gareth P Seaward, MB, BCh, MSc, Principal Investigator — Mt.Sinai Hospital, University of Toronto, Canada
Locations (1):
- Mt. Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Oepkes D, Seaward PG, Vandenbussche FP, Windrim R, Kingdom J, Beyene J, Kanhai HH, Ohlsson A, Ryan G; DIAMOND Study Group. Doppler ultrasonography versus amniocentesis to predict fetal anemia. N Engl J Med. 2006 Jul 13;355(2):156-64. doi: 10.1056/NEJMoa052855. PMID 16837679